CLINICAL TRIAL: NCT04338880
Title: The Associations of High Academic Performance With Childhood Ametropia Prevalence and Myopia Progression
Brief Title: Academic Performance and Refractive Error
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Sun Yat-sen University
Other Study IDs: CCPMOH2016-China-0901
Record Dates: First submitted 2020-04-07; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Refractive errors constitute the leading cause of visual disability worldwide and that myopia progresses dramatically when students reach school age. Studies from different countries have reported inconsistent associations between educational outcomes and refractive errors. Therefore, our study aimed to assess the associations of high academic performance with ametropia prevalence and myopia progression in Chinese schoolchildren base on a multicohort observational design.

ELIGIBILITY:
Inclusion Criteria:

* schoolchildren in the 1st to 9th grades

Exclusion Criteria:

* schoolchildren unwilling to participate
* had a history of wearing rigid contact lenses, medical treatment or diseases that could cause poor vision or negatively affect the academic outcomes
* with unreliable auto-refraction values

Ages: 6 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: A prospective multicohort observational study of schoolchildren who studied in the 1st to 9th grades was performed.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
the changes of spherical equivalent refractive (RSE) | up to 3 years
  A multi-linear regression was used.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China